CLINICAL TRIAL: NCT06924567
Title: The Accuracy of CT-based Implant Movement for the Evaluation of Cup and Stem Stability, When Plain Radiography is Not Conclusive for Loosening, in Patients Scheduled for Revision Hip Arthroplasty. A Multicenter Study
Brief Title: Radiographic Stability of Hip Prosthesis Prior to Revision Surgery
Acronym: MULTICIMA
Status: Not yet recruiting | Type: Observational
Sponsor: Georgios Tsikandylakis, MD PhD (Other)
Collaborators: Sectra AB, Sweden (Unknown)
Responsible Party: Sponsor-Investigator, Georgios Tsikandylakis, MD PhD, MD, PhD, Sahlgrenska University Hospital
Organization: Sahlgrenska University Hospital (Other)
Other Study IDs: 284803
Record Dates: First submitted 2025-04-05; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Loosening, Prosthesis; Hip Arthropathy
Keywords: implant stabilty; THA; radiographic evaluation; IMA; Implant Movement Analysis; Revision THA
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Study group: Patients with painful THA, scheduled for reviision hip arthoplasty, with no signs of obvious implant loosening in either the cup or the stem.
  Interventions: Diagnostic Test: Implant motion provocation CT

INTERVENTIONS:
Diagnostic Test: Implant motion provocation CT — Implant Movement Analysis. A low dose CT scan is performed with the hip fixed in external rotation. Then another low dose CT scan is performed with the hip fixed in internal rotation.The CT scans are then overimposed to each other and implant motion in relation to host bone is visualized,

SUMMARY:
The goal of this validation study is to compare the preoperative implant stability, assessed by Implant Movement Analysis (IMA), provocation dual CT scans, with the intraoperative stability evaluation in revision hip arthoplasty. The main question it aims to answer is:

Does IMA reflect the intraoperative clinical evaluation of implant stability? Participants scheduled for revision hip arthoplasty will undergo IMA preoperativelly in addition to rutine clinical work up. During revision arthoplasty, a surgeon blinded to the IMA results will assess clinically the stability of the hip prosthesis. IMA will be compared with the intraoperative findings to assess IMAs sensitivity and specificity

ELIGIBILITY:
Inclusion criteria: 600 consecutive patients scheduled for revision THA due to aseptic loosening, in whom, one component has no convincing loosening signs, based on the preoperative plain radiographs and clinical assessment by the attending surgeon. The radiographs should be not older than 8 weeks prior to surgery.

Exclusion criteria:

Both cup and stem have been preoperatively evaluated as loose by the attending surgeon, based on the preoperative plain radiographs.

Instability with repeating dislocation of the THA Non-aseptic revision surgery, based on preoperative work up. Participants are excluded after inclusion if revision surgery is cancelled.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a painful total hip arthoplasty that are scheduled for revision hip arthoplasty due to suspected prosthesis loosening. At least one implant component (either cup or stem) should not have any obvious signs of loosening. Only the implant component with no obvious signs of loosening will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Cup and stem stability | within 2 months month
  The stability of the cup and the stem is evaluated:
  1. Preoperatively with IMA as binary outcome (loose/not loose).
  2. Intraoperatively by the surgeon as binary outcome (loose/notloose).

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Malchau, MD, PhD, Study Chair — Sahlgrenska University Hospital; Georgios Tsikandylakis, Principal Investigator — Sahlgrenska University Hospital
Locations (4):
- Sweden (4):
  - Sahlgrenska University Hospital, Gothenburg
  - Hässleholm Hospital, Hässleholm
  - Danderyd Hospital, Stockholm
  - Akademiska University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Olivecrona H, Olivecrona L, Weidenhielm L, Noz ME, Kardos J, Maguire GQ Jr, Zeleznik MP, Aspelin P. A new technique for diagnosis of acetabular cup loosening using computed tomography: preliminary experience in 10 patients. Acta Orthop. 2008 Jun;79(3):346-53. doi: 10.1080/17453670710015247. PMID 18622838
- [Background] Lovera D, Sandberg O, Mohaddes M, Gyllensten H. Cost-effectiveness of implant movement analysis in aseptic loosening after hip replacement: a health-economic model. Cost Eff Resour Alloc. 2023 Nov 20;21(1):88. doi: 10.1186/s12962-023-00498-w. PMID 37986000
- [Background] Sandberg O, Carlsson S, Harbom E, Cappelen V, Tholen S, Olivecrona H, Wretenberg P. Inducible displacement CT increases the diagnostic accuracy of aseptic loosening in primary total hip arthroplasty. Acta Orthop. 2022 Oct 31;93:831-836. doi: 10.2340/17453674.2022.5240. PMID 36314542